CLINICAL TRIAL: NCT00854048
Title: The Performance of Nellcor OxiMax N-560 and Masimo SET Radical Pulse Oximeters in Pediatric Patients With Low Oxygen Saturation Levels
Brief Title: The Performance of Pulse Oximeters in Pediatric Patients With Low Oxygen Saturation Levels
Status: Completed | Type: Observational
Sponsor: Ulf Borg (Industry)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor-Investigator, Ulf Borg, Director Clinical Science, Medtronic - MITG
Organization: Medtronic - MITG (Industry)
Other Study IDs: M112
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Cardiopulmonary Bypass
Keywords: Pediatric; Oxygen Saturation; Cardiopulmonary bypass

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Evaluate pulse oximeters with children after cardiopulmonary by-pass under low Oxygen conditions.

ELIGIBILITY:
Inclusion Criteria:

* Include pediatric patients with a baseline Sa02 < 90% and no contraindications to using an adhesive sensor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric patients after cardiopulmonary by-pass in the PICU.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xu Feng, MD, Principal Investigator — Children's Hospital Congqing Medical University
Locations (1):
- Chidren's Hospital, Chongqing University of Medical Sciences, Chongqing Municipality, China